CLINICAL TRIAL: NCT02667392
Title: Biofeedback to Increase Propulsion During Walking After Stroke
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N2051-P
Record Dates: First submitted 2016-01-19; First posted 2016-01-28 (Estimated); Results first posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Stroke
Keywords: Stroke; Gait; Walking; Rehabilitation; Exercise; Exercise Therapy; Physical Therapy Modalities; Exercise Movement Techniques
MeSH Terms: conditions — Stroke; Motor Activity | interventions — Biofeedback, Psychology

STUDY DESIGN:
Intervention Model Description: Parallel: participants are assigned to one of two or more groups in parallel for the duration of the study.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Biofeedback Group (Experimental): Participants will wear a pressure-sensitive insole inside the shoe of their paretic limb. An auditory tone will sound when participants have provided sufficient load to active the pressure-sensitive in-sole.
  Interventions: Procedure: Gait Training with Biofeedback
- Verbal Feedback Group (Active Comparator): Participants will receive verbal feedback from a physical therapist regarding the amount of loading they are exerting on their paretic limb.
  Interventions: Procedure: Gait Training with Verbal Feedback

INTERVENTIONS:
Procedure: Gait Training with Biofeedback — Intervention (12, 60-minute sessions, 3X/week for four weeks) will occur in an outpatient research setting. Participants will be supervised by a licensed physical therapist and wear a gait belt during all activities. The therapist will choose from a standardized bank of gait activities, suitable to each participant's ability level. The goal for total walking time for each session will be 50 minutes: 5, 10-minute bouts with a 2-minute rest between bouts. This is the typical length and intensity of outpatient rehabilitation sessions for ambulatory patients discharged from inpatient rehabilitation.
  Biofeedback Group: Biofeedback (external-focus feedback) will be provided as an adjuvant to therapist-provided feedback during the intervention. Participants will be instructed that a tone will sound when they "push off with their (paretic) leg to swing it forward" when the participant-specific pre-programmed threshold is exceeded.
  Arms: Biofeedback Group
Procedure: Gait Training with Verbal Feedback — Intervention (12, 60-minute sessions, 3X/week for four weeks) will occur in an outpatient research setting. Participants will be supervised by a licensed physical therapist and wear a gait belt during all activities. The therapist will choose from a standardized bank of gait activities, suitable to each participant's ability level. The goal for total walking time for each session will be 50 minutes: 5, 10-minute bouts with a 2-minute rest between bouts. This is the typical length and intensity of outpatient rehabilitation sessions for ambulatory patients discharged from inpatient rehabilitation.
  Verbal Feedback Group: Therapist-provided internal-focus feedback ("directed towards components of body movement") will be used to instruct participants on achieving and/or maintaining appropriate movement patterns that contribute to propulsion generation.
  Arms: Verbal Feedback Group

SUMMARY:
Approximately 15,000 Veterans are hospitalized for stroke each year with new cases costing an estimated $111 million for acute inpatient, $75 million for post-acute inpatient, and $88 million for follow-up care over 6 months post-stroke. Rehabilitation of walking ability contributes to these costs. To "walk again" is the number one stated goal for Veterans who have had a stroke. Teaching patients post-stroke to use their weak leg while they are regaining walking function and to not compensate by over-using their strong leg is necessary to restore safe, efficient walking ability. This project will determine if providing biofeedback (an audible tone) from pressure-sensitive shoe insole sensors, that encourage use of the weaker leg during walking training, in addition to therapists' feedback, will help Veterans regain use of their weak leg, improve their endurance and improve their balance when walking in challenging environments.

DETAILED DESCRIPTION:
Background/Purpose: Approximately 15,000 Veterans are hospitalized for stroke each year. Impairments of motor control and the subsequent functional limitations in ambulation are the most common manifestations and regaining the ability to walk is the number one stated goal of Veteran stroke survivors. Forward propulsion of the body's center of mass is a cardinal feature of gait that depends on the generation of appropriate anterior-posterior ground reaction forces. Decreased propulsive force generation by the paretic limb of stroke survivors has been identified through both simulation and cross-sectional studies as a major contributor to walking dysfunction. Extrinsic verbal feedback from a therapist is the standard approach used during gait retraining to improve propulsion generation. However, this key component of gait is not directly observable by therapists and patients are often unable to sense propulsion generation due to impaired intrinsic feedback, specifically deficits in somatosensation and proprioception, hindering recovery of paretic propulsion and compromising walking function. The objective of this study is to provide preliminary evidence that biofeedback as an adjuvant to therapists' verbal feedback will improve propulsion and enhance walking function for Veterans post-stroke.

Subjects: Thirty individuals > 6-months post-stroke will participate. Additional study criteria include: 1) Ambulation of household distances without physical assistance to advance or support the paretic leg; 2) Unilateral leg paresis confirmed by a score of < 32 on the Fugl-Meyer Motor Assessment; 3) Step length asymmetry (paretic > non-paretic step length); 4) Ambulation without an assistive or orthotic device.

Methods: Participants will be randomized to either an experimental group that will train with propulsion biofeedback from commercially available pressure-sensitive insole sensors (Biofeedback group; n=15) or a control group that will train with standard therapist-provided verbal feedback alone (Standard group; n=15). The 12 session (3X/week for 4 weeks) gait training intervention will be delivered by a physical therapist-led team. For participants in the Biofeedback group, prior to the first intervention session, the baseline amount of pressure exerted by the paretic forefoot during late stance will be determined. The insole area underlying the forefoot will then be calibrated to produce a tone when pressure exceeds 5% of this baseline pressure. This threshold will be progressively increased at regular intervals throughout the intervention period to ensure participants are training at their challenge-point to improve propulsion of the paretic limb. An insole of similar thickness will be worn in the shoe of the non-paretic leg for symmetry and comfort but will not produce a tone during the intervention. Those in the Standard group will not wear insoles during intervention but will receive verbal feedback alone regarding propulsion of the paretic limb during gait training. Therapist-provided verbal feedback will be used to instruct participants on achieving and/or maintaining appropriate movement patterns that contribute to propulsion generation. For both groups, the therapist will choose from a standardized bank of gait activities, suitable to each participant's ability level. The goal for total walking time for each session will be 50 minutes: 5, 10-minute bouts with a 2-minute rest between each bout.

Outcome Measures: Paretic limb propulsion is the primary outcome measure. Secondary measures include the Six Minute Walk Test, Functional Gait Assessment, Fall Self-Efficacy, temporal-distance gait measures and gait kinematics, all of which will be measured pre- and post-intervention.

Data Analysis Plan: Descriptive statistics will be provided for all outcome measures. To identify the effect of the intervention, differences between the pre- and post-training assessment within each group (i.e. change scores) will be calculated. To test the hypotheses, the investigators will apply independent sample t-tests to the change scores of the Biofeedback and Standard group. Hypothesis testing will be conducted at a two-sided p < 0.05 level.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stroke
* > 6 months < 5 years post-stroke onset
* Medically stable
* 18-80 years of age
* Impaired lower extremity sensation confirmed by a score of < 12 on the Fugl-Meyer Sensory Assessment,20
* Community-dwelling
* Step length asymmetry (paretic step length > non-paretic step length)

  * this asymmetry has been determined to be correlated with minimal propulsive force of the paretic leg4
* Unilateral lower extremity paresis confirmed by a score of < 32 on the Fugl-Meyer Motor Assessment,20
* Able to ambulate without an orthotic device
* Able to ambulate without an assistive device
* Ambulation of household distances without physical assistance to advance or support paretic lower extremity

Exclusion Criteria:

* Presence of a neurological condition other than stroke
* Pain upon ambulation
* Receiving physical therapy services for mobility and/or gait
* Severe arthritis or orthopedic problems that limit passive ranges of motion

  * knee flexion contracture of -10 , knee flexion range of motion (ROM) < 90
  * hip flexion contracture > 25
  * ankle plantar flexion contracture > 15

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2019-09-16 (Actual); Study Completion 2019-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dorian Kay Rose, PhD MS BS, Principal Investigator — North Florida/South Georgia Veterans Health System, Gainesville, FL
Locations (1):
- North Florida/South Georgia Veterans Health System, Gainesville, FL, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled between October 2017 and August 2019. Study site was the Brain Rehabilitation Research Center at the Malcom Randall Veterans Affairs Medical Center - akin to an "outpatient" site.
Pre-assignment Details: The original study design was to have two arms: 1) Biofeedback arm, 2) Verbal feedback arm.
  Secondary to construction of the laboratory space where the study was to take place and delayed human resources hiring of study personnel, recruitment for this study was delayed. It was determined that the most prudent course of action would be to conduct a single-arm study with all participants being assigned to the biofeedback arm.
Groups:
- Biofeedback Group: Participants will wear a pressure-sensitive insole inside the shoe of their paretic limb. An auditory tone will sound when participants have provided sufficient load to active the pressure-sensitive in-sole.
  Gait Training with Biofeedback: Intervention (12, 60-minute sessions, 3 times/week for four weeks) will occur in an outpatient research setting. Participants will be supervised by a licensed physical therapist and wear a gait belt during all activities. The therapist will choose from a standardized bank of gait activities, suitable to each participant's ability level. The goal for total walking time for each session will be 50 minutes: 5, 10-minute bouts with a 2-minute rest between bouts. This is the typical length and intensity of outpatient rehabilitation sessions for ambulatory patients discharged from inpatient rehabilitation.
  Biofeedback Group: Biofeedback (external-focus feedback) will be provided as an adjuvant to therapist-provided feedback during the intervention. Participants will be instructed that a tone will sound when they "push off with their (paretic) leg to swing it forward" when the participant-specific pre-programmed threshold is exceeded.
Period: Overall Study
Arm/Group | Biofeedback Group
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The original study design was to have two arms: 1) Biofeedback arm, 2) Verbal feedback arm.
  Secondary to construction of the laboratory space where the study was to take place and delayed human resources hiring of study personnel, recruitment for this study was delayed. It was determined that the most prudent course of action to study the efficacy of this experimental biofeedback intervention would be to conduct a single-arm study with all participants being assigned to the biofeedback arm.
Arm/Group | Biofeedback Group
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.0 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Time Since Stroke Onset [Mean (Standard Deviation); unit: months] | 40.4 (29.1)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Forward Propulsion of the Paretic Limb From Pre- to Post-intervention
Description: The propulsive impulse will be derived from the time integral of the positive anterior-posterior ground reaction force for the paretic leg normalized to Body Weight.
Time Frame: Pre-intervention (prior to 1st intervention session) and Post-intervention (after the final (12th intervention session), approximately 4 weeks after entering the study.
Population: as for baseline characteristics
Measure: Mean (Standard Error); unit: Newtons . seconds/Body Weight
Arm/Group | Biofeedback Group
Number analyzed (Participants) | 11
Newtons . seconds/Body Weight | 0.00 (.017)
Statistical Analysis 1: Comparison: Biofeedback Group; Test type: Other; p = 0.77, t-test, 2 sided — a priori threshold for statistical significance set at p < 0.05

2. Secondary Outcome: Change From Baseline in Peak Hip Flexion Range of Motion, in Degrees, of the Paretic Leg From Pre- to Post-intervention
Description: Hip motion data will be acquired using a modified Helen Hayes marker set with rigid clusters on the pelvis and each thigh and reflective markers at the greater trochanter and the lateral condyle of the femur. The angle formed between the rigid cluster on the pelvis and the lateral condyle of the femur will be recorded at 100 Hz using a 12 camera motion capture system. The peak value from 10 gait cycles was averaged to obtain an average peak value.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Mean (Standard Error); unit: degrees
Arm/Group | Biofeedback Group
Number analyzed (Participants) | 11
degrees | 1.5 (2.9)
Statistical Analysis 1: Comparison: Biofeedback Group; Test type: Other; p = 0.61, t-test, 2 sided — a priori threshold for statistical significance set at p < 0.05

3. Secondary Outcome: Change From Baseline in Stride Time From Pre to Post-intervention.
Description: Data will be acquired while walking across a GAITRite instrumented walkway.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Mean (Standard Error); unit: Seconds
Arm/Group | Biofeedback Group
Number analyzed (Participants) | 11
Seconds | 0.1 (0)
Statistical Analysis 1: Comparison: Biofeedback Group; Test type: Other; p = 0.28, t-test, 2 sided — a priori threshold for statistical significance set at p < 0.05

4. Secondary Outcome: Change From Baseline in Distance Covered During the Six Minute Walk Test From Pre- to Post-intervention
Description: Participants will walk for a total of six minutes at their comfortable walking speed and the total distance will be recorded.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Mean (Standard Error); unit: Meters
Arm/Group | Biofeedback Group
Number analyzed (Participants) | 11
Meters | 44 (11.4)
Statistical Analysis 1: Comparison: Biofeedback Group; Test type: Other; p = 0.002, t-test, 2 sided — a priori threshold for statistical significance set at p < 0.05

5. Secondary Outcome: Change From Baseline in the Functional Gait Assessment Score From Pre- to Post-intervention
Description: Ten item gait and balance test during which participants walk forwards, backwards, ascend/descend stairs, walk with head turning and step over obstacles. Score ranges from 0-30 with a larger number indicative of a better outcome. Each item is scored on a 0-4 scale with a lower number representing greater impairment. The individual score on each of the ten items are summed for a total score with a larger number indicative of a better outcome.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Biofeedback Group
Number analyzed (Participants) | 11
score on a scale | 2.1 (0.8)
Statistical Analysis 1: Comparison: Biofeedback Group; Test type: Other; p = 0.02, t-test, 2 sided — a priori threshold for statistical significance set at p < 0.05

6. Secondary Outcome: Change From Baseline in the Modified Falls Efficacy Scale From Pre- to Post-intervention
Description: Fourteen item questionnaire designed to measure self-perceived fear of falling during task performance. Score range is between 0-10 with a higher score indicative of a better outcome
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Biofeedback Group
Number analyzed (Participants) | 11
score on a scale | 0.8 (0.4)
Statistical Analysis 1: Comparison: Biofeedback Group; Test type: Other; p = 0.03, t-test, 2 sided — a priori threshold for statistical significance set at p < 0.05

7. Secondary Outcome: Change From Baseline in Paretic Limb Step Time From Pre- to Post-intervention.
Description: Footfall of both limbs will be acquired while participants walk across a pressure sensitive instrumented walkway (GAITRite). From these footballs paretic step time will be calculated.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Mean (Standard Error); unit: Seconds
Arm/Group | Biofeedback Group
Number analyzed (Participants) | 11
Seconds | .04 (.07)
Statistical Analysis 1: Comparison: Biofeedback Group; Test type: Other; p = 0.55, t-test, 2 sided — a priori threshold for statistical significance set at p < 0.05

8. Secondary Outcome: Change From Baseline in Paretic Limb Stride Length From Pre to Post-intervention.
Description: Footfalls from both limbs will be acquired as participant walks across a pressure-sensitive instrumented walkway (GAITRite). From these footfalls will be used to calculate paretic limb stride length.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Mean (Standard Error); unit: Meters
Arm/Group | Biofeedback Group
Number analyzed (Participants) | 11
Meters | .05 (.02)
Statistical Analysis 1: Comparison: Biofeedback Group; Test type: Other — a priori threshold for statistical significance set at p < 0.05; p = 0.0089, t-test, 2 sided

9. Secondary Outcome: Change From Baseline in Paretic Limb Step Length From Pre to Post-intervention.
Description: Footfalls from both limbs will be acquired as participant walks across a pressure-sensitive instrumented walkway (GAITRite). From these footfalls will be used to calculate paretic limb step length.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Mean (Standard Error); unit: Meters
Arm/Group | Biofeedback Group
Number analyzed (Participants) | 11
Meters | .01 (.02)
Statistical Analysis 1: Comparison: Biofeedback Group; Test type: Other — a priori threshold for statistical significance set at p < 0.05; p = 0.73, t-test, 2 sided

10. Secondary Outcome: Change From Baseline in Paretic Limb Step Width From Pre to Post-intervention.
Description: Footfalls from both limbs will be acquired as participant walks across a pressure-sensitive instrumented walkway (GAITRite). From these footfalls will be used to calculate paretic limb step width.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Mean (Standard Error); unit: Meters
Arm/Group | Biofeedback Group
Number analyzed (Participants) | 11
Meters | 0.0 (0.0)
Statistical Analysis 1: Comparison: Biofeedback Group; Test type: Other — a priori threshold for statistical significance set at p < 0.05; p = 0.81, t-test, 2 sided

11. Secondary Outcome: Change From Baseline in Gait Speed From Pre to Post-intervention.
Description: Data will be acquired while participants walk across a pressure-sensitive 14 meter instrumented walkway (Brand Name: GAITRite).
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Mean (Standard Error); unit: meters/second
Arm/Group | Biofeedback Group
Number analyzed (Participants) | 11
meters/second | 0.14 (.07)
Statistical Analysis 1: Comparison: Biofeedback Group; Test type: Other; p = 0.02, t-test, 2 sided — a priori threshold for statistical significance set at p < 0.05

ADVERSE EVENTS:
Time Frame: Each participant was enrolled in the study for six weeks. Adverse Event data was collected for the six weeks participants were enrolled in the study.
Description: The original study design was to have two arms: 1) Biofeedback arm, 2) Verbal feedback arm.
  Secondary to construction of the laboratory space where the study was to take place and delayed human resources hiring of study personnel, recruitment for this study was delayed. It was determined that the most prudent course of action to study the efficacy of this experimental biofeedback intervention would be to conduct a single-arm study with all participants being assigned to the biofeedback arm.
Arm/Group | Biofeedback Group
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-08): https://cdn.clinicaltrials.gov/large-docs/92/NCT02667392/Prot_SAP_000.pdf